CLINICAL TRIAL: NCT02969616
Title: A Prospective, Post Market, Multi-center, Open Label, Non-Randomized Clinical Study of the Efficacy of Using Trinity ELITE in Lumbar Fusion Surgery
Brief Title: Trinity Elite in Lumbar Fusion
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1504TEPL
Record Dates: First submitted 2016-11-15; First posted 2016-11-21 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Degenerative Disc Disease
Keywords: lumbar, fusion, DDD, Trinity Elite
MeSH Terms: conditions — Intervertebral Disc Degeneration; Dowling-Degos Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Trinity Elite — cell based allograft

SUMMARY:
This prospective, post-market, open label clinical study is designed to examine the lumbar fusion rate at 24 months post operative in subjects who have undergone a lumbar fusion surgery using Trinity Elite with or without local bone.

DETAILED DESCRIPTION:
The study is a prospective, post-market, open label clinical study. Up to 10 sites across the United States, with a minimum enrollment of 120 subjects study-wide, will be enrolling subjects. The primary objective of this study is to measure the lumbar fusion rate in subjects at 24 months when lumbar arthrodesis is performed using Trinity Elite with or without local bone. Surgical approach (PLF, TLIF,ALIF, XLIF, etc.) is according to the physician's discretion, but must comply with FDA approved/cleared indication for use and labeling. The primary endpoints are radiographic evidence of fusion and the absence of serious adverse events attributable to Trinity ELITE. The secondary objectives of this study are to measure the clinical and economic outcomes when posterolateral arthrodesis is performed using Trinity Elite and/or local bone with supplemental pedicle screw fixation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years of age (≥ 18 years) or older at the time of consent.
2. Subject must have a documented diagnosis of DDD. DDD is defined by back and/or radicular pain with degeneration of the disc as confirmed by medical history, physical examination, and radiographic studies that may include CT, MRI, plain X-ray film, discography, myelography, etc. with one or more of the following findings:

   * Instability as defined by >3mm translation or >5 degrees angulation
   * Osteophyte formation of facet joints or vertebral endplates
   * Decreased disc height, on average by >2mm, but dependent upon the spinal level
   * Scarring/thickening of ligamentum flavum, annulus fibrosis, or facet joint capsule
   * Herniated nucleus pulposus
   * Facet joint degeneration/changes; and/or
   * Vacuum phenomenon
3. Subject may have up to a Grade 2 Spondylolisthesis of the lumbar spine with clinical manifestations of one or more of the following phenomena:

   * Radiculopathy
   * Sensory deficit
   * Motor weakness
   * Reflex changes
4. Subject must require lumbar arthrodesis at 1-4 contiguous levels (L1-S1) for a PLF approach and 1-2 contiguous levels for an interbody approach.
5. Subject must have been unresponsive to conservative care for at least 6 months prior to fusion surgery.

7. Subject must agree not to use electromagnetic adjuncts to enhance bone fusion during the course of the study 8. Subject must be willing and able to sign an informed consent document. 9. Subject must be willing and able to return for all follow-up visits, agree to participate in postoperative clinical and radiographic evaluations and comply with the required study regimen.

Exclusion Criteria:

1. Subject is under 18 years of age (<18) at the time of consent
2. Subject has had prior lumbar spine fusion surgery at any level
3. Subject has greater than grade 2 spondylolisthesis of the lumbar spine
4. Subject is currently undergoing treatment for malignancy or has undergone treatment for malignancy in the past 5 years (benign skin cancer is permitted)
5. Subject is pregnant or nursing or planning to become pregnant during the two years (24 months) following arthrodesis
6. Subject has an active local or systemic infection or is undergoing adjunctive treatment for local or systemic infection
7. Subject requires supplemental interbody arthrodesis.
8. Subject has an allergy to DMSO.
9. Subject is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age >= 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-09; Primary Completion 2022-02 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
lumbar fusion by CT scan following arthrodesis using Trinity Elite | 24 months
  CT scan of the lumbar vertebral column will be used to determine the fusion status of the spine after Trinity Elite was used in the lateral gutters and in the facet joints. The number of bridging bony cortices will be recorded by blinded reviewers and tabulated. The data will be reported as n
number of participants with treatment related adverse events | 24 months
  AEs collected on an ongoing basis, reviewed by the Investigators and medical monitor

CONTACTS AND LOCATIONS:
Overall Officials: Alan Daniels, MD, Principal Investigator — Brown University; Daniel Park, MD, Principal Investigator — Beaumont Hospital; Fernando Techy, MD, Principal Investigator — ClinTech Center for Spine Health

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lansford T, Park DK, Wind JJ, Nunley P, Peppers TA, Russo A, Hassanzadeh H, Sembrano J, Yoo J, Sales J. High Lumbar Spinal Fusion Rates Using Cellular Bone Allograft Irrespective of Surgical Approach. Int J Spine Surg. 2024 Sep 12;18(4):355-364. doi: 10.14444/8612. PMID 39054302
- [Derived] Russo A, Park DK, Lansford T, Nunley P, Peppers TA, Wind JJ, Hassanzadeh H, Sembrano J, Yoo J, Sales J. Impact of surgical risk factors for non-union on lumbar spinal fusion outcomes using cellular bone allograft at 24-months follow-up. BMC Musculoskelet Disord. 2024 May 3;25(1):351. doi: 10.1186/s12891-024-07456-4. PMID 38702654
- [Derived] Park DK, Wind JJ, Lansford T, Nunley P, Peppers TA, Russo A, Hassanzadeh H, Sembrano J, Yoo J, Sales J. Twenty-four-month interim results from a prospective, single-arm clinical trial evaluating the performance and safety of cellular bone allograft in patients undergoing lumbar spinal fusion. BMC Musculoskelet Disord. 2023 Nov 17;24(1):895. doi: 10.1186/s12891-023-06996-5. PMID 37978378